CLINICAL TRIAL: NCT05750498
Title: Autoimmune Liver Disease Network for Kids (A-LiNK): Using Patient Data to Transform Care and Improve Outcomes for Children, Adolescents, and Young Adults With Autoimmune Liver Disease
Brief Title: A-LiNK: Improving Outcomes in Autoimmune Liver Disease
Acronym: ALINK
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-1019 A-LiNK Prospective
Record Dates: First submitted 2023-02-13; First posted 2023-03-01 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Autoimmune Hepatitis; Primary Sclerosing Cholangitis
Keywords: Pediatrics; Autoimmune Hepatitis; Primary Sclerosing Cholangitis; Autoimmune Sclerosing Cholangitis; Chronic Liver Disease; End-stage Liver Disease; Clinical Registry; Research Registry; Quality Improvement; Outcomes Research; Comparative Effectiveness Research; Patient Reported Outcomes; Health Services Research
MeSH Terms: conditions — Hepatitis, Autoimmune; Cholangitis, Sclerosing; End Stage Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children and adolescents with Autoimmune Liver Disease: Pediatric patients with a diagnosis of autoimmune hepatitis, or primary sclerosing cholangitis.
  Interventions: Other: No interventions

INTERVENTIONS:
Other: No interventions — There are no interventions

SUMMARY:
The Autoimmune Liver disease Network for Kids (A-LiNK) is a multi-institutional group with the mission to deliver the best care to kids with pediatric autoimmune liver disease (AILD).

This study will establish a shared clinical registry and a learning health network for the participating sites focusing on collecting and transmitting clinical measurement data, information about processes, and participation in an improvement collaborative.

Pediatric Autoimmune Hepatitis (AIH) and Primary Sclerosing Cholangitis (PSC), represent a spectrum of AILD which present unique diagnostic and therapeutic challenges.A lack of accepted guidelines for disease monitoring or symptom management results in wide treatment variation with liver transplants indicated in refractory, progressive disease.

The aims of A-LiNK are to:

1.) Create a learning health network focused on patient-centered outcomes research characterized by transparent sharing among centers, common priorities, and feasible plans for implementing new practices; 2) shift from traditional investigator-driven study to a patient and family-centered approach, and 3.) improve clinical outcomes and quality of life for pediatric AILD patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of autoimmune hepatitis (AIH)
* Clinical diagnosis of primary sclerosing cholangitis (PSC)
* Clinical diagnosis of autoimmune sclerosing cholangitis (ASC)

Exclusion Criteria:

• History of liver transplant

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with a clinical diagnosis of Autoimmune Hepatitis (AIH), Primary Sclerosing Cholangitis (PSC), and Autoimmune Sclerosing Cholangitis (ASC).
  Patient recruitment will be conducted by the care centers participating in the registry.
  This also includes the recruitment of Spanish and other language-speaking patients.
  Participants who are enrolled in ImproveCareNow and who are eligible for A-LiNK will be separately consented to this study.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2022-04-28 (Actual); Primary Completion 2032-12-31 (Estimated); Study Completion 2033-06-30 (Estimated)

PRIMARY OUTCOMES:
Baseline disease characteristics in the population | 2034
Disease relapse and biochemical remission rates | 2034
  Biochemical remission = transaminases (ALT/AST) within the upper limit of normal for age
Complications of disease | 2034
  Including ascites, esophageal variceal bleeding, cholangitis, hepatic encephalopathy, listed for liver transplant, hepatocellular carcinoma, or cholangiocarcinoma
Side-effects of steroids | 2034
  Including hypertension, diabetes mellitus, low bone mineral density, glaucoma, cataract, overweight, obesity
Pediatric Quality of Life Inventory (PedsQL 4.0) Generic Core Scales Short Form 15 | 2034
  Health-related quality of life
Racial and ethnic disparities | 2034

CONTACTS AND LOCATIONS:
Overall Officials: Amy E Taylor, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (8):
- United States (8):
  - Stanford University, Palo Alto, California
  - Riley Children's Health, Indianapolis, Indiana
  - St. Louis Children's Hospital, St Louis, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
To expand the possibilities for conducting outcomes research beyond the A-LiNK network of investigators, data will be shared, following an internal review process, with qualified investigators external to the network who are employed at, or affiliated with, institutions that are interested in conducting health services or comparative effectiveness research. Following a merit review and legal agreement, a de-identified data set will be shared with investigators following a workflow documented in the data-sharing procedure.
  To share data with investigators in and outside the network, the A-LiNK Leadership Committee will ensure that any requests that constitute research involving human subjects have received appropriate institutional review board (IRB) review and approval prior the sharing of data.